CLINICAL TRIAL: NCT02314143
Title: Phase II Biomarker Study Evaluating The Upfront Combination Of BRAF Inhibitor Dabrafenib With MEK Inhibitor Trametinib Versus The Combination After Eight Weeks Of Monotherapy With Dabrafenib Or Trametinib In Patients With Metastatic And Unresectable Stage III Or IV Melanoma Harbouring An Activating BRAF Mutation
Brief Title: Phase II Biomarker Study Comparing the Combination of BRAF Inhibitor Dabrafenib With MEK Inhibitor Trametinib Versus the Combination After Monotherapy With Dabrafenib or Trametinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to slow enrollment and limited numbers of viable tissue samples.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 116613
Record Dates: First submitted 2013-09-25; First posted 2014-12-11 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-09

CONDITIONS: Melanoma
Keywords: dabrafenib; MEK; trametinib; BRAF; melanoma; Oncology
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dabrafenib followed by combination therapy (Experimental): Eligible subjects will receive dabrafenib 150 milligrams (mg) twice a day (BID) continuously during 8 weeks of monotherapy treatment followed by the combination of trametinib 2 mg once daily with dabrafenib 150 mg BID until disease progression, death or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Trametinib followed by combination therapy (Experimental): Eligible subjects will receive trametinib 2 mg per day continuously during 8 weeks of monotherapy treatment followed by the combination of trametinib 2 mg once daily with dabrafenib 150 mg BID until disease progression, death or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Combination therapy (Experimental): Eligible subjects will receive trametinib 2 mg per day plus dabrafenib 150 mg BID continuously until disease progression, death or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib will be provided as 50 mg and 75 mg capsules.
Drug: Trametinib — Trametinib study medication will be provided as 0.5 mg and 2.0 mg tablets.

SUMMARY:
This is a three-arm, open-label, randomised Phase II study to evaluate whether the different sequencing of dabrafenib and trametinib monotherapies and the upfront combination has an impact on translational or clinical activity in subjects with BRAF mutant metastatic unresectable stage IIIc or IV melanoma. Both dabrafenib and trametinib have demonstrated clinical activity as monotherapies and in combination in BRAF-mutant melanoma. However, duration of responses seem to be limited due to acquired drug resistance. The goal of this protocol is to study the sequential effects of BRAF and MEK inhibition on skin, blood and tumour biomarkers and to study the correlation between biomarkers and response to treatment and intrapatient toxicity. Approximately 54 eligible subjects will be randomised in the ratio of 1:1:1 to one of the three treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Participant with signed written informed consent;
* Participants of age >=18 years;
* Participants with histologically confirmed cutaneous melanoma that is either Stage IIIc (unresectable) or Stage IV (metastatic) (according to American Joint Committee on Cancer [AJCC] staging 7th edition).
* BRAF (proto-oncogene B-Raf) V600E/K mutation-positive confirmed by a local laboratory.
* Accessible melanoma tumours for biopsies (locally advanced primary melanoma or metastases)
* Measurable disease according to Response Evaluation Criteria in Solid Tumours (RECIST 1.1) on not biopsied lesions.
* All prior anti-cancer treatment-related toxicities (except alopecia) must be <= Grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.0) at the time of randomisation.
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomisation and agree to use effective contraception, throughout the treatment period, and for 4 months after the last dose of study treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Adequate baseline organ function as defined : absolute neutrophil count >= 1.2 × 109/Liters (L); Haemoglobin >= 9 grams(g)/Deciliter (dL); Platelet count >= 75 x 109/L; prothrombin time(PT)/ international normalized ratio (INR) and partial thromboplastin time (PTT) <= 1.5 x Upper limit of normal (ULN); Albumin >= 2.5 g/dL; Total bilirubin- <= 1.5 x ULN; aspartate aminotransferase(AST) and alanine transaminase (ALT) <= 2.5 x ULN; Calculated creatinine clearance >=50 mL/min; Left Ventricular Ejection fraction (LVEF) >= Lower limit of normal (LLN) by Echocardiogram (ECHO)

Exclusion Criteria:

* Prior treatment with a BRAF or MEK inhibitor
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to randomisation and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to randomisation.
* Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to randomisation
* Current use of a prohibited medication.
* Refusal of tumour and skin biopsies.
* History of another malignancy.
* Any serious and/or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the participant's safety, obtaining informed consent, or compliance with study procedures.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which will be allowed).
* A history of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Brain metastases are excluded unless: All known lesions were previously treated with surgery or stereotactic surgery (whole-brain radiation is not allowed unless given after definitive treatment with surgery or stereotactic surgery), OR Brain lesion(s), if still present, must be confirmed stable (i.e., no increase in lesion size) for >= 12 weeks prior to randomisation (stability must be confirmed with two consecutive magnetic resonance image (MRI) or computed tomography (CT) scans with contrast, AND Asymptomatic with no corticosteroid requirements for >= 4 weeks prior to randomisation, AND No enzyme inducing anticonvulsants for >= 4 weeks prior to randomisation.
* A history or evidence of cardiovascular risk including any of the following: LVEF < LLN; A QT interval corrected for heart rate using the Bazett's formula (QTcB) >= 480 milliseconds (msec); A history or evidence of current clinically significant uncontrolled arrhythmias; Exception: Participants with atrial fibrillation controlled for > 30 days prior to randomisation are eligible; A history (within 6 months prior to randomisation) of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty; A history or evidence of current >= Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines; Treatment refractory hypertension defined as a blood pressure of systolic > 140 millimetres of mercury (mmHg) and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy; Participants with intra-cardiac defibrillators or permanent pacemakers; Known cardiac metastases; Abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (Participants with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Participants with moderate valvular thickening should not be entered on study.
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including: Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR such as: Evidence of new optic disc cupping; Evidence of new visual field defects on automated perimetry; Intraocular pressure >21 mmHg as measured by tonography.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* Pregnant or lactating females
* Interstitial lung disease or pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Villejuif
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open label, randomized, phase II study to compare the combination of dabrafenib with trametinib versus the combination after eight weeks of monotherapy with dabrafenib or trametinib in metastatic and unresectable stage III or IV melanoma. The study was terminated early due to slow enrollment and limited numbers of viable tissue samples.
Pre-assignment Details: This study was planned to enroll 54 participants randomized in 1:1:1 ratio into the three treatment arms; dabrafenib followed by combination therapy, trametinib followed by combination therapy and only combination therapy. The study was early terminated with 48 participants enrolled.
Groups:
- Dabrafenib Followed by Combination Therapy: Eligible participants received dabrafenib 150 milligrams (mg) twice a day (BID) continuously during 8 weeks of monotherapy treatment followed by the combination of trametinib 2 mg once daily with dabrafenib 150 mg BID until disease progression, death or unacceptable toxicity.
- Trametinib Followed by Combination Therapy: Eligible participants received trametinib 2 mg per day continuously during 8 weeks of monotherapy treatment followed by the combination of trametinib 2 mg once daily with dabrafenib 150 mg BID until disease progression, death or unacceptable toxicity.
- Combination Therapy: Eligible participants received trametinib 2 mg per day plus dabrafenib 150 mg BID continuously until disease progression, death or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Started | 16 | 16 | 16
Completed | 8 | 6 | 7
Not Completed | 8 | 10 | 9
Not completed — Adverse Event | 0 | 6 | 4
Not completed — Other (Study Closed/Terminated) | 5 | 3 | 4
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (16.43) | 56.5 (11.77) | 58.9 (13.55) | 57.4 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 21
  Male | 9 | 8 | 10 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-South East Asian Heritage | 0 | 1 | 0 | 1
  White - White/Caucasian/European | 16 | 15 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Percentage Change From Baseline in Extracellular Signal-regulated Kinase (ERK) Phosphorylation (p-ERK) H Score From Week 0 to Week 2
Description: Intra-tumoral expression levels of ERK measured using immunohistochemistry methods. The H score value ranged from 0 to a maximum score of 300 (strongest expression) was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0 [no staining], 1+ [weak staining], 2+ [medium staining] and 3+ [strongest staining]). Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. Percentage change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplied by 100. The data has been presented for combination therapy calculated from Week 0 to Week 2. The analysis was based on the biomarker Population which included all participants with biopsy performed at screening and at least once during treatment.
Time Frame: Baseline (Week 0) and up to 2 weeks
Population: Biomarker Population. Only those participants with data available at specific time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 5
Participants
  Any Increase or No Changes | 2
  Any Decrease up to 80 percent | 1
  Any Decrease > 80 percent | 2

2. Primary Outcome: Number of Participants With Percentage Change in p-ERK H Score From Week 8 to Week 10
Description: Intra-tumoral expression levels of ERK were measured using immunohistochemistry methods. The H score value ranged from 0 to a maximum score of 300 (strongest expression) was derived by summing the percentages of cells staining at each intensity multiplied by the weighted intensity of staining (0 [no staining], 1+ [weak staining], 2+ [medium staining] and 3+ [strongest staining]). Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. Percentage change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplied by 100. The data has been presented for dabrafenib followed by combination therapy and trametinib followed by combination therapy, calculated from Week 8 to Week 10.
Time Frame: Week 8 and up to 10 weeks
Population: Biomarker Population. Only those participants with data available at specific time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy
Number analyzed (Participants) | 1 | 3
Participants
  Any Increase or No Changes | 1 | 1
  Any Decrease up to 80 percent | 0 | 1
  Any Decrease > 80 percent | 0 | 1

3. Secondary Outcome: Number of Participants With Overall Response Rate (ORR)
Description: Clinical response was evaluated by ORR, which was defined as the number of participants with a confirmed or an unconfirmed complete response (CR) or partial response (PR) at any time per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. CR was defined as disappearance of all target lesions. PR was defined as at least a 30 percent decrease in the sum of the diameters of target lesions. Number of participants with ORR (CR+PR) has been presented. The analysis was based on the Intent-to-Treat Population (ITT) which included all the randomized participants whether or not randomized treatment was administered.
Time Frame: Up to 3.2 years
Population: Intent-to-Treat Population (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants | 11 | 13 | 11
Statistical Analysis 1: Comparison: Dabrafenib Followed by Combination Therapy vs Combination Therapy; Test type: Other; p = 1.0000, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.224 to 4.459] — The odds ratio for dabrafenib followed by combination therapy versus combination therapy has been presented
Statistical Analysis 2: Comparison: Trametinib Followed by Combination Therapy vs Combination Therapy; Test type: Other; p = 0.4216, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.970, 95% CI 2-sided [0.382 to 10.166] — The odds ratio for trametinib followed by combination therapy versus combination therapy has been presented

4. Secondary Outcome: Number of Participants With Change in Vital Signs From Baseline
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and heat rate (HR) were measured. Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus the Baseline value. The number of participants with heart rate "decrease to < 60" and "increase to >100" have been presented. For SBP and DBP, "any grade increase" have been presented. Any grade increase in SBP, including grade 0 (<120), grade 1 (120-139), grade 2 (140-159), grade 3 (>=160) and DBP including grade 0 (<80), grade 1 (80-89), grade 2 (90-99), grade 3 (>=100) have been presented. The analysis was based on the Safety Population which included all participants who received at least one dose of randomized treatment and was based on the actual treatment received. Only those participants available at specified time point were analyzed (represented by n=x in category titles).
Time Frame: Baseline and up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  HR; Week 4; Decrease to <60; n=15,16,16: number analyzed (Participants) | 15 | 16 | 16
  HR; Week 4; Decrease to <60; n=15,16,16 | 1 | 3 | 3
  HR; Week 4; Increase to >100; n=15,16,16: number analyzed (Participants) | 15 | 16 | 16
  HR; Week 4; Increase to >100; n=15,16,16 | 1 | 0 | 0
  HR; Week 8; Decrease to <60; n=16,16,14: number analyzed (Participants) | 16 | 16 | 14
  HR; Week 8; Decrease to <60; n=16,16,14 | 1 | 2 | 2
  HR; Week 8; Increase to >100; n=16,16,14: number analyzed (Participants) | 16 | 16 | 14
  HR; Week 8; Increase to >100; n=16,16,14 | 2 | 0 | 0
  HR; Week 12; Decrease to <60; n=16,16,13: number analyzed (Participants) | 16 | 16 | 13
  HR; Week 12; Decrease to <60; n=16,16,13 | 2 | 1 | 2
  HR; Week 12; Increase to >100; n=16,16,13: number analyzed (Participants) | 16 | 16 | 13
  HR; Week 12; Increase to >100; n=16,16,13 | 0 | 0 | 0
  HR; Week 16; Decrease to <60; n=14,16,13: number analyzed (Participants) | 14 | 16 | 13
  HR; Week 16; Decrease to <60; n=14,16,13 | 0 | 0 | 2
  HR; Week 16; Increase to >100; n=14,16,13: number analyzed (Participants) | 14 | 16 | 13
  HR; Week 16; Increase to >100; n=14,16,13 | 0 | 0 | 0
  HR; Week 20; Decrease to <60; n=11,15,13: number analyzed (Participants) | 11 | 15 | 13
  HR; Week 20; Decrease to <60; n=11,15,13 | 0 | 1 | 1
  HR; Week 20; Increase to >100; n=11,15,13: number analyzed (Participants) | 11 | 15 | 13
  HR; Week 20; Increase to >100; n=11,15,13 | 1 | 1 | 0
  HR; Week 24; Decrease to <60; n=12,14,13: number analyzed (Participants) | 12 | 14 | 13
  HR; Week 24; Decrease to <60; n=12,14,13 | 1 | 2 | 2
  HR; Week 24; Increase to >100; n=12,14,13: number analyzed (Participants) | 12 | 14 | 13
  HR; Week 24; Increase to >100; n=12,14,13 | 1 | 2 | 0
  HR; Week 28; Decrease to <60; n=8,12,7: number analyzed (Participants) | 8 | 12 | 7
  HR; Week 28; Decrease to <60; n=8,12,7 | 2 | 2 | 2
  HR; Week 28; Increase to >100; n=8,12,7: number analyzed (Participants) | 8 | 12 | 7
  HR; Week 28; Increase to >100; n=8,12,7 | 1 | 0 | 0
  HR; Week 32; Decrease to <60; n=7,11,8: number analyzed (Participants) | 7 | 11 | 8
  HR; Week 32; Decrease to <60; n=7,11,8 | 1 | 0 | 0
  HR; Week 32; Increase to >100; n=7,11,8: number analyzed (Participants) | 7 | 11 | 8
  HR; Week 32; Increase to >100; n=7,11,8 | 1 | 0 | 0
  HR; Week 36; Decrease to <60; n=5,11,8: number analyzed (Participants) | 5 | 11 | 8
  HR; Week 36; Decrease to <60; n=5,11,8 | 2 | 0 | 1
  HR; Week 36; Increase to >100; n=5,11,8: number analyzed (Participants) | 5 | 11 | 8
  HR; Week 36; Increase to >100; n=5,11,8 | 0 | 0 | 1
  HR; Week 40; Decrease to <60; n=6,11,7: number analyzed (Participants) | 6 | 11 | 7
  HR; Week 40; Decrease to <60; n=6,11,7 | 1 | 1 | 0
  HR; Week 40; Increase to >100; n=6,11,7: number analyzed (Participants) | 6 | 11 | 7
  HR; Week 40; Increase to >100; n=6,11,7 | 0 | 0 | 0
  HR; Week 44; Decrease to <60; n=5,5,4: number analyzed (Participants) | 5 | 5 | 4
  HR; Week 44; Decrease to <60; n=5,5,4 | 1 | 0 | 0
  HR; Week 44; Increase to >100; n=5,5,4: number analyzed (Participants) | 5 | 5 | 4
  HR; Week 44; Increase to >100; n=5,5,4 | 1 | 0 | 1
  HR; Week 48; Decrease to <60; n=5,4,4: number analyzed (Participants) | 5 | 4 | 4
  HR; Week 48; Decrease to <60; n=5,4,4 | 1 | 0 | 1
  HR; Week 48; Increase to >100; n=5,4,4: number analyzed (Participants) | 5 | 4 | 4
  HR; Week 48; Increase to >100; n=5,4,4 | 0 | 0 | 1
  HR; Week 52; Decrease to <60; n=4,3,4: number analyzed (Participants) | 4 | 3 | 4
  HR; Week 52; Decrease to <60; n=4,3,4 | 0 | 0 | 0
  HR; Week 52; Increase to >100; n=4,3,4: number analyzed (Participants) | 4 | 3 | 4
  HR; Week 52; Increase to >100; n=4,3,4 | 0 | 0 | 1
  HR; Week 56; Decrease to <60; n=4,3,4: number analyzed (Participants) | 4 | 3 | 4
  HR; Week 56; Decrease to <60; n=4,3,4 | 1 | 0 | 3
  HR; Week 56; Increase to >100; n=4,3,4: number analyzed (Participants) | 4 | 3 | 4
  HR; Week 56; Increase to >100; n=4,3,4 | 0 | 0 | 0
  HR; Week 60; Decrease to <60; n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  HR; Week 60; Decrease to <60; n=3,3,4 | 1 | 1 | 1
  HR; Week 60; Increase to >100; n=3,3,4: number analyzed (Participants) | 3 | 3 | 4
  HR; Week 60; Increase to >100; n=3,3,4 | 0 | 0 | 0
  HR; Week 64; Decrease to <60; n=3,3,3: number analyzed (Participants) | 3 | 3 | 3
  HR; Week 64; Decrease to <60; n=3,3,3 | 1 | 0 | 0
  HR; Week 64; Increase to >100; n=3,3,3: number analyzed (Participants) | 3 | 3 | 3
  HR; Week 64; Increase to >100; n=3,3,3 | 0 | 0 | 0
  HR; Week 68; Decrease to <60; n=4,2,2: number analyzed (Participants) | 4 | 2 | 2
  HR; Week 68; Decrease to <60; n=4,2,2 | 1 | 0 | 2
  HR; Week 68; Increase to >100; n=4,2,2: number analyzed (Participants) | 4 | 2 | 2
  HR; Week 68; Increase to >100; n=4,2,2 | 0 | 0 | 0
  HR; Week 72; Decrease to <60; n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  HR; Week 72; Decrease to <60; n=3,2,2 | 0 | 0 | 0
  HR; Week 72; Increase to >100; n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  HR; Week 72; Increase to >100; n=3,2,2 | 0 | 0 | 0
  HR; Week 76; Decrease to <60; n=4,1,2: number analyzed (Participants) | 4 | 1 | 2
  HR; Week 76; Decrease to <60; n=4,1,2 | 1 | 0 | 0
  HR; Week 76; Increase to >100; n=4,1,2: number analyzed (Participants) | 4 | 1 | 2
  HR; Week 76; Increase to >100; n=4,1,2 | 0 | 0 | 1
  HR; Week 80; Decrease to <60; n=3,1,2: number analyzed (Participants) | 3 | 1 | 2
  HR; Week 80; Decrease to <60; n=3,1,2 | 1 | 0 | 0
  HR; Week 80; Increase to >100; n=3,1,2: number analyzed (Participants) | 3 | 1 | 2
  HR; Week 80; Increase to >100; n=3,1,2 | 0 | 0 | 0
  HR; Week 84; Decrease to <60; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 84; Decrease to <60; n=3,1,1 | 0 | 0 | 0
  HR; Week 84; Increase to >100; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 84; Increase to >100; n=3,1,1 | 0 | 0 | 0
  HR; Week 88; Decrease to <60; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 88; Decrease to <60; n=3,1,1 | 1 | 0 | 0
  HR; Week 88; Increase to >100; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 88; Increase to >100; n=3,1,1 | 0 | 0 | 0
  HR; Week 92; Decrease to <60; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 92; Decrease to <60; n=3,1,1 | 1 | 0 | 0
  HR; Week 92; Increase to >100; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 92; Increase to >100; n=3,1,1 | 0 | 0 | 0
  HR; Week 96; Decrease to <60; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 96; Decrease to <60; n=3,1,1 | 1 | 0 | 0
  HR; Week 96; Increase to >100; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 96; Increase to >100; n=3,1,1 | 0 | 0 | 0
  HR; Week 100; Decrease to <60; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 100; Decrease to <60; n=3,1,1 | 0 | 0 | 0
  HR; Week 100; Increase to >100; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 100; Increase to >100; n=3,1,1 | 0 | 0 | 0
  HR; Week 104; Decrease to <60; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 104; Decrease to <60; n=3,1,1 | 0 | 0 | 0
  HR; Week 104; Increase to >100; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  HR; Week 104; Increase to >100; n=3,1,1 | 0 | 0 | 0
  HR; Week 108; Decrease to <60; n=2,0,1: number analyzed (Participants) | 2 | 0 | 1
  HR; Week 108; Decrease to <60; n=2,0,1 | 1 |  | 0
  HR; Week 108; Increase to >100; n=2,0,1: number analyzed (Participants) | 2 | 0 | 1
  HR; Week 108; Increase to >100; n=2,0,1 | 0 |  | 0
  HR; Week 112; Decrease to <60; n=2,0,0: number analyzed (Participants) | 2 | 0 | 0
  HR; Week 112; Decrease to <60; n=2,0,0 | 1 |  |
  HR; Week 112; Increase to >100; n=2, 0,0: number analyzed (Participants) | 2 | 0 | 0
  HR; Week 112; Increase to >100; n=2, 0,0 | 0 |  |
  HR; Week 116; Decrease to <60; n=1, 0,0: number analyzed (Participants) | 1 | 0 | 0
  HR; Week 116; Decrease to <60; n=1, 0,0 | 0 |  |
  HR; Week 116; Increase to >100; n=1, 0,0: number analyzed (Participants) | 1 | 0 | 0
  HR; Week 116; Increase to >100; n=1, 0,0 | 0 |  |
  HR; Week 120; Decrease to <60; n=1, 0,0: number analyzed (Participants) | 1 | 0 | 0
  HR; Week 120; Decrease to <60; n=1, 0,0 | 0 |  |
  HR; Week 120; Increase to >100; n=1, 0,0: number analyzed (Participants) | 1 | 0 | 0
  HR; Week 120; Increase to >100; n=1, 0,0 | 0 |  |
  HR; Week 124; Decrease to <60; n=1, 0,0: number analyzed (Participants) | 1 | 0 | 0
  HR; Week 124; Decrease to <60; n=1, 0,0 | 0 |  |
  HR; Week 124; Increase to >100; n=1, 0,0: number analyzed (Participants) | 1 | 0 | 0
  HR; Week 124; Increase to >100; n=1, 0,0 | 0 |  |
  SBP; Week 4; Any grade increase; n=15,16,16: number analyzed (Participants) | 15 | 16 | 16
  SBP; Week 4; Any grade increase; n=15,16,16 | 1 | 8 | 4
  SBP; Week 8; Any grade increase; n=16,16,14: number analyzed (Participants) | 16 | 16 | 14
  SBP; Week 8; Any grade increase; n=16,16,14 | 3 | 5 | 4
  SBP; Week 12; Any grade increase; n=16,16,13: number analyzed (Participants) | 16 | 16 | 13
  SBP; Week 12; Any grade increase; n=16,16,13 | 3 | 5 | 2
  SBP; Week 16; Any grade increase; n=14,16,13: number analyzed (Participants) | 14 | 16 | 13
  SBP; Week 16; Any grade increase; n=14,16,13 | 4 | 3 | 2
  SBP; Week 20; Any grade increase; n=11,15, 13: number analyzed (Participants) | 11 | 15 | 13
  SBP; Week 20; Any grade increase; n=11,15, 13 | 2 | 3 | 1
  SBP; Week 24; Any grade increase; n=12, 14,13: number analyzed (Participants) | 12 | 14 | 13
  SBP; Week 24; Any grade increase; n=12, 14,13 | 2 | 3 | 2
  SBP; Week 28; Any grade increase; n=8, 12,7: number analyzed (Participants) | 8 | 12 | 7
  SBP; Week 28; Any grade increase; n=8, 12,7 | 2 | 0 | 0
  SBP; Week 32; Any grade increase; n=7,11, 8: number analyzed (Participants) | 7 | 11 | 8
  SBP; Week 32; Any grade increase; n=7,11, 8 | 2 | 3 | 2
  SBP; Week 36; Any grade increase; n=5, 11, 8: number analyzed (Participants) | 5 | 11 | 8
  SBP; Week 36; Any grade increase; n=5, 11, 8 | 3 | 3 | 1
  SBP; Week 40; Any grade increase; n=6,11, 7: number analyzed (Participants) | 6 | 11 | 7
  SBP; Week 40; Any grade increase; n=6,11, 7 | 1 | 4 | 2
  SBP; Week 44; Any grade increase; n=5, 5, 4: number analyzed (Participants) | 5 | 5 | 4
  SBP; Week 44; Any grade increase; n=5, 5, 4 | 2 | 0 | 0
  SBP; Week 48; Any grade increase; n=5,4, 4: number analyzed (Participants) | 5 | 4 | 4
  SBP; Week 48; Any grade increase; n=5,4, 4 | 1 | 1 | 0
  SBP; Week 52; Any grade increase; n=4,3, 4: number analyzed (Participants) | 4 | 3 | 4
  SBP; Week 52; Any grade increase; n=4,3, 4 | 1 | 0 | 0
  SBP; Week 56; Any grade increase; n=4, 3, 4: number analyzed (Participants) | 4 | 3 | 4
  SBP; Week 56; Any grade increase; n=4, 3, 4 | 0 | 0 | 0
  SBP; Week 60; Any grade increase; n=3, 2, 4: number analyzed (Participants) | 3 | 2 | 4
  SBP; Week 60; Any grade increase; n=3, 2, 4 | 1 | 1 | 0
  SBP; Week 64; Any grade increase; n=3, 3, 3: number analyzed (Participants) | 3 | 3 | 3
  SBP; Week 64; Any grade increase; n=3, 3, 3 | 1 | 0 | 0
  SBP; Week 68; Any grade increase; n=4,2, 2: number analyzed (Participants) | 4 | 2 | 2
  SBP; Week 68; Any grade increase; n=4,2, 2 | 2 | 0 | 0
  SBP; Week 72; Any grade increase; n=3,2, 2: number analyzed (Participants) | 3 | 2 | 2
  SBP; Week 72; Any grade increase; n=3,2, 2 | 1 | 0 | 0
  SBP; Week 76; Any grade increase; n=4, 1, 2: number analyzed (Participants) | 4 | 1 | 2
  SBP; Week 76; Any grade increase; n=4, 1, 2 | 2 | 0 | 0
  SBP; Week 80; Any grade increase; n=3, 1, 2: number analyzed (Participants) | 3 | 1 | 2
  SBP; Week 80; Any grade increase; n=3, 1, 2 | 2 | 0 | 0
  SBP; Week 84; Any grade increase; n=3, 1,1: number analyzed (Participants) | 3 | 1 | 1
  SBP; Week 84; Any grade increase; n=3, 1,1 | 2 | 0 | 0
  SBP; Week 88; Any grade increase; n=3, 1,1: number analyzed (Participants) | 3 | 1 | 1
  SBP; Week 88; Any grade increase; n=3, 1,1 | 0 | 0 | 0
  SBP; Week 92; Any grade increase; n=3, 1, 1: number analyzed (Participants) | 3 | 1 | 1
  SBP; Week 92; Any grade increase; n=3, 1, 1 | 2 | 0 | 0
  SBP; Week 96; Any grade increase; n=3,1, 1: number analyzed (Participants) | 3 | 1 | 1
  SBP; Week 96; Any grade increase; n=3,1, 1 | 2 | 1 | 0
  SBP; Week 100; Any grade increase; n=3, 1, 1: number analyzed (Participants) | 3 | 1 | 1
  SBP; Week 100; Any grade increase; n=3, 1, 1 | 0 | 0 | 0
  SBP; Week 104; Any grade increase; n=3, 1, 1: number analyzed (Participants) | 3 | 1 | 1
  SBP; Week 104; Any grade increase; n=3, 1, 1 | 1 | 0 | 0
  SBP; Week 108; Any grade increase; n=2,0, 1: number analyzed (Participants) | 2 | 0 | 1
  SBP; Week 108; Any grade increase; n=2,0, 1 | 1 |  | 0
  SBP; Week 112; Any grade increase; n=2, 0, 0: number analyzed (Participants) | 2 | 0 | 0
  SBP; Week 112; Any grade increase; n=2, 0, 0 | 0 |  |
  SBP; Week 116; Any grade increase; n=1, 0, 0: number analyzed (Participants) | 1 | 0 | 0
  SBP; Week 116; Any grade increase; n=1, 0, 0 | 0 |  |
  SBP; Week 120; Any grade increase; n=1, 0, 0: number analyzed (Participants) | 1 | 0 | 0
  SBP; Week 120; Any grade increase; n=1, 0, 0 | 0 |  |
  SBP; Week 124; Any grade increase; n=1, 0, 0: number analyzed (Participants) | 1 | 0 | 0
  SBP; Week 124; Any grade increase; n=1, 0, 0 | 0 |  |
  DBP; Week 4; Any grade increase; n=15, 16, 16: number analyzed (Participants) | 15 | 16 | 16
  DBP; Week 4; Any grade increase; n=15, 16, 16 | 2 | 10 | 5
  DBP; Week 8; Any grade increase; n=16, 16,14: number analyzed (Participants) | 16 | 16 | 14
  DBP; Week 8; Any grade increase; n=16, 16,14 | 4 | 8 | 3
  DBP; Week 12; Any grade increase; n=16, 16, 13: number analyzed (Participants) | 16 | 16 | 13
  DBP; Week 12; Any grade increase; n=16, 16, 13 | 4 | 4 | 2
  DBP; Week 16; Any grade increase; n=14, 16,13: number analyzed (Participants) | 14 | 16 | 13
  DBP; Week 16; Any grade increase; n=14, 16,13 | 5 | 5 | 3
  DBP; Week 20; Any grade increase; n=11, 15,13: number analyzed (Participants) | 11 | 15 | 13
  DBP; Week 20; Any grade increase; n=11, 15,13 | 4 | 5 | 2
  DBP; Week 24; Any grade increase; n=12, 14,13: number analyzed (Participants) | 12 | 14 | 13
  DBP; Week 24; Any grade increase; n=12, 14,13 | 3 | 3 | 1
  DBP; Week 28; Any grade increase; n=8, 12,7: number analyzed (Participants) | 8 | 12 | 7
  DBP; Week 28; Any grade increase; n=8, 12,7 | 1 | 2 | 0
  DBP; Week 32; Any grade increase; n=7, 11,8: number analyzed (Participants) | 7 | 11 | 8
  DBP; Week 32; Any grade increase; n=7, 11,8 | 2 | 3 | 1
  DBP; Week 36; Any grade increase; n=5, 11,8: number analyzed (Participants) | 5 | 11 | 8
  DBP; Week 36; Any grade increase; n=5, 11,8 | 2 | 1 | 2
  DBP; Week 40; Any grade increase; n=6, 11,7: number analyzed (Participants) | 6 | 11 | 7
  DBP; Week 40; Any grade increase; n=6, 11,7 | 1 | 1 | 1
  DBP; Week 44; Any grade increase; n=5, 5,4: number analyzed (Participants) | 5 | 5 | 4
  DBP; Week 44; Any grade increase; n=5, 5,4 | 4 | 1 | 2
  DBP; Week 48; Any grade increase; n=5, 4,4: number analyzed (Participants) | 5 | 4 | 4
  DBP; Week 48; Any grade increase; n=5, 4,4 | 2 | 1 | 2
  DBP; Week 52; Any grade increase; n=4,3,4: number analyzed (Participants) | 4 | 3 | 4
  DBP; Week 52; Any grade increase; n=4,3,4 | 2 | 0 | 0
  DBP; Week 56; Any grade increase; n=4,3,4: number analyzed (Participants) | 4 | 3 | 4
  DBP; Week 56; Any grade increase; n=4,3,4 | 1 | 1 | 0
  DBP; Week 60; Any grade increase; n=3,2,4: number analyzed (Participants) | 3 | 2 | 4
  DBP; Week 60; Any grade increase; n=3,2,4 | 2 | 0 | 0
  DBP; Week 64; Any grade increase; n=3,3, 3: number analyzed (Participants) | 3 | 3 | 3
  DBP; Week 64; Any grade increase; n=3,3, 3 | 1 | 0 | 1
  DBP; Week 68; Any grade increase; n=4,2, 2: number analyzed (Participants) | 4 | 2 | 2
  DBP; Week 68; Any grade increase; n=4,2, 2 | 2 | 0 | 1
  DBP; Week 72; Any grade increase; n=3,2,2: number analyzed (Participants) | 3 | 2 | 2
  DBP; Week 72; Any grade increase; n=3,2,2 | 1 | 0 | 1
  DBP; Week 76; Any grade increase; n=4,1,2: number analyzed (Participants) | 4 | 1 | 2
  DBP; Week 76; Any grade increase; n=4,1,2 | 2 | 0 | 1
  DBP; Week 80; Any grade increase; n=3,1,2: number analyzed (Participants) | 3 | 1 | 2
  DBP; Week 80; Any grade increase; n=3,1,2 | 1 | 0 | 1
  DBP; Week 84; Any grade increase; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  DBP; Week 84; Any grade increase; n=3,1,1 | 1 | 0 | 0
  DBP; Week 88; Any grade increase; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  DBP; Week 88; Any grade increase; n=3,1,1 | 1 | 0 | 0
  DBP; Week 92; Any grade increase; n=3, 1,1: number analyzed (Participants) | 3 | 1 | 1
  DBP; Week 92; Any grade increase; n=3, 1,1 | 1 | 0 | 1
  DBP; Week 96; Any grade increase; n=3, 1,1: number analyzed (Participants) | 3 | 1 | 1
  DBP; Week 96; Any grade increase; n=3, 1,1 | 2 | 0 | 1
  DBP; Week 100; Any grade increase; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  DBP; Week 100; Any grade increase; n=3,1,1 | 1 | 0 | 0
  DBP; Week 104; Any grade increase; n=3,1,1: number analyzed (Participants) | 3 | 1 | 1
  DBP; Week 104; Any grade increase; n=3,1,1 | 1 | 0 | 1
  DBP; Week 108; Any grade increase; n=2,0,1: number analyzed (Participants) | 2 | 0 | 1
  DBP; Week 108; Any grade increase; n=2,0,1 | 1 |  | 0
  DBP; Week 112; Any grade increase; n=2,0,0: number analyzed (Participants) | 2 | 0 | 0
  DBP; Week 112; Any grade increase; n=2,0,0 | 0 |  |
  DBP; Week 116; Any grade increase; n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  DBP; Week 116; Any grade increase; n=1,0,0 | 0 |  |
  DBP; Week 120; Any grade increase; n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  DBP; Week 120; Any grade increase; n=1,0,0 | 0 |  |
  DBP; Week 124; Any grade increase; n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  DBP; Week 124; Any grade increase; n=1,0,0 | 0 |  |

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings Undergoing Physical Examinations
Description: Complete physical examination included assessments of eyes, neurological and cardiovascular systems, lungs, abdomen, and any other areas with signs and symptoms of disease, and of the head, neck, ears, nose, mouth, throat, thyroid, lymph nodes, extremities, and a full skin exam to assess cutaneous malignancies and proliferative skin diseases. This analysis was planned but data was not captured in the database. Abnormal changes were captured as adverse events if they were clinically significant.
Time Frame: Up to 3.2 years
Population: Safety Population. This analysis was planned but data was not captured in the database.
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Change in Eastern Cooperative Oncology Group (ECOG) Performance Status Scores From Baseline
Description: The ECOG scale of performance status describes the level of functioning of participants in terms of their ability to care for themselves, daily activity, and physical ability. The ECOG performance was recorded as per ECOG performance status grades ranging from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead). Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The Baseline performance status of participants with respect to worst-case on-therapy performance status has been presented.
Time Frame: Baseline and up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  0 to 0 | 5 | 5 | 6
  0 to 1 | 0 | 0 | 1
  0 to 2 | 0 | 0 | 0
  0 to 3 | 0 | 0 | 0
  0 to 4-5 | 0 | 0 | 0
  1 to 0 | 6 | 10 | 5
  1 to 1 | 3 | 1 | 2
  1 to 2 | 0 | 0 | 0
  1 to 3 | 0 | 0 | 0
  1 to 4-5 | 0 | 0 | 0
  2 to 0 | 0 | 0 | 0
  2 to 1 | 2 | 0 | 2
  2 to 2 | 0 | 0 | 0
  2 to 3 | 0 | 0 | 0
  2 to 4-5 | 0 | 0 | 0
  3 to 0 | 0 | 0 | 0
  3 to 1 | 0 | 0 | 0
  3 to 2 | 0 | 0 | 0
  3 to 3 | 0 | 0 | 0
  3 to 4-5 | 0 | 0 | 0
  4-5 to 0 | 0 | 0 | 0
  4-5 to 1 | 0 | 0 | 0
  4-5 to 2 | 0 | 0 | 0
  4-5 to 3 | 0 | 0 | 0
  4-5 to 4-5 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECG) Findings
Description: Single measurements of 12-lead ECGs were obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, corrected QT interval (QTc), Bazett's Corrected QT interval (QTcB), Friderica's Corrected QT interval (QTcF). Number of participants with abnormal ECG findings (Abnormal - Not Clinically Significant and Abnormal - Clinically Significant ) at any time post-Baseline visit have been presented.
Time Frame: Up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  Abnormal - Not Clinically Significant | 9 | 10 | 9
  Abnormal - Clinically Significant | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Absolute Change in Left Ventricular Ejection Fraction From Baseline
Description: Echocardiograms (ECHO) was performed to assess cardiac ejection fraction and cardiac valve morphology. Baseline was defined as the most recent non-missing value prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The worst-case on-therapy value has been presented.
Time Frame: Baseline and up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  No Change Or Any Increase | 11 | 14 | 11
  >0-<10 Decrease | 4 | 2 | 3
  >=10 Decrease And >= Lower limit of Normal (Lln) | 1 | 0 | 2

9. Secondary Outcome: Number of Participants With Change in Clinical Chemistry Parameters From Baseline
Description: Blood samples were collected for evaluation of clinical chemistry parameters including sodium, potassium, calcium, albumin, total protein, blood urea nitrogen (BUN), creatinine, lactate dehydrogenase (LDH), gamma-glutamyl transpeptidase (GCT), phosphate, C-reactive protein (CRP), hypercalcemia, hyperkalemia, hypernatremia, hypocalcemia, hypokalemia, hyponatremia, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin, direct bilirubin and estimated creatinine clearance (CRTCE). Baseline was defined as the most recent non-missing value from a central laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The worst-case on therapy value for number of participants with any grade increase in clinical chemistry parameters for has been presented. Only those participants available at specified time point were analyzed (represented by n=x in category titles).
Time Frame: Baseline and up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  ALT; n=16,16,16 | 3 | 13 | 9
  Albumin; n=16,16,16 | 2 | 5 | 2
  Alkaline phosphatase; n=16,16,16 | 5 | 10 | 4
  AST; n=16,16,16 | 8 | 15 | 12
  Bilirubin; n=16,16,16 | 0 | 2 | 0
  CRP;n=12,12,13: number analyzed (Participants) | 12 | 12 | 13
  CRP;n=12,12,13 | 0 | 0 | 0
  Creatinine; n=16,16,16 | 0 | 0 | 0
  Direct bilirubin; n=4,6,3: number analyzed (Participants) | 4 | 6 | 3
  Direct bilirubin; n=4,6,3 | 0 | 0 | 0
  GCT; n=16,16,16 | 6 | 12 | 5
  Hypercalcemia; n=16,16,16 | 0 | 0 | 0
  Hyperkalemia; n=16,16,16 | 1 | 4 | 0
  Hypernatremia; n=16,16,16 | 3 | 4 | 1
  Hypocalcemia; n=16,16,16 | 7 | 7 | 4
  Hypokalemia; n=16,16,16 | 1 | 4 | 3
  Hyponatremia; n=16,16,16 | 7 | 7 | 5
  LDH; 16,16,15: number analyzed (Participants) | 16 | 16 | 15
  LDH; 16,16,15 | 0 | 0 | 0
  Phosphate; n=16,16,16 | 10 | 6 | 4
  Protein; n=16,16,16 | 0 | 0 | 0
  Urea; n=15,15,16: number analyzed (Participants) | 15 | 15 | 16
  Urea; n=15,15,16 | 0 | 0 | 0
  CRTCE; n=5,2,5: number analyzed (Participants) | 5 | 2 | 5
  CRTCE; n=5,2,5 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Change in Hematology Parameters From Baseline
Description: Blood samples were collected for evaluation of hematology parameters including hemoglobin, white blood cell (WBC), platelet count, basophils, eosinophils, lymphocytes, monocytes, total neutrophils, lymphocytopenia and lymphocytosis. Baseline was defined as the most recent non-missing value from a central laboratory prior to the first dose of study treatment. Change from Baseline was defined as any visit value minus Baseline value. The worst-case on therapy value for number of participants with any grade increase in hematology parameters for has been presented.
Time Frame: Baseline and up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  Basophils | 0 | 0 | 0
  Eosinophils | 0 | 0 | 0
  Hemoglobin | 4 | 6 | 4
  Leukocytes | 5 | 9 | 10
  Monocytes | 0 | 0 | 0
  Neutrophils | 6 | 9 | 9
  Platelets | 2 | 5 | 3
  Lymphocytopenia | 8 | 6 | 6
  Lymphocytosis | 2 | 0 | 0

11. Secondary Outcome: Number of Participants With Incidence of Squamous Cell Carcinoma and Keratoacanthoma
Description: The safety profile of dabrafenib and trametinib in monotherapy as well as in combination therapy was characterized by determining the number of participants with incidence of squamous cell carcinoma and keratoacanthoma.
Time Frame: Up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants | 1 | 0 | 0

12. Secondary Outcome: Number of Participants With On-treatment Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function.
Time Frame: Up to 3.2 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 16 | 16 | 16
Participants
  Any Non-SAE | 16 | 16 | 15
  Any SAE | 8 | 7 | 4

13. Secondary Outcome: Plasma Pharmacokinetic Concentration of Trametinib
Description: Blood samples were collected for pharmacokinetic analysis of trametinib at indicated time points. Pharmacokinetic analysis was performed using standard non-compartmental method.
Time Frame: 4 to 8 hours post-dose at Weeks 2, 8 and 10
Population: Biomarker Population. Only those participants with data available at specific time point were analyzed (represented by n=x in category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 13 | 14 | 15
Nanograms per milliliter
  WEEK 2 ; 4 to 8 HOURS POST-DOSE; n= 12, 14,13: number analyzed (Participants) | 12 | 14 | 13
  WEEK 2 ; 4 to 8 HOURS POST-DOSE; n= 12, 14,13 | 1.4 (4.99) | 14.6 (5.15) | 16.3 (5.73)
  WEEK 8 ; 4 to 8 HOURS POST-DOSE; n=12, 12, 10: number analyzed (Participants) | 12 | 12 | 10
  WEEK 8 ; 4 to 8 HOURS POST-DOSE; n=12, 12, 10 | 0.6 (2.06) | 12.9 (8.82) | 13.8 (6.46)
  WEEK 10 ; 4 to 8 HOURS POST-DOSE; n=13, 13, 11: number analyzed (Participants) | 13 | 13 | 11
  WEEK 10 ; 4 to 8 HOURS POST-DOSE; n=13, 13, 11 | 10.5 (5.33) | 8.8 (7.50) | 14.7 (6.66)

14. Secondary Outcome: Plasma Pharmacokinetic Concentration of Dabrafenib
Description: Blood samples were collected for pharmacokinetic analysis of Dabrafenib at indicated time points. Pharmacokinetic analysis was performed using standard non-compartmental method.
Time Frame: 4 to 8 hours post-dose at Weeks 2, 8 and 10
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
Number analyzed (Participants) | 13 | 14 | 15
Nanograms per milliliter
  WEEK 2 ; 4 to 8 HOURS POST-DOSE; n= 12, 14,13: number analyzed (Participants) | 12 | 14 | 13
  WEEK 2 ; 4 to 8 HOURS POST-DOSE; n= 12, 14,13 | 219.7 (545.46) | 0.0 (0.00) | 438.1 (487.26)
  WEEK 8 ; 4 to 8 HOURS POST-DOSE; n=12, 12, 10: number analyzed (Participants) | 12 | 12 | 10
  WEEK 8 ; 4 to 8 HOURS POST-DOSE; n=12, 12, 10 | 259.1 (669.60) | 0.0 (0.00) | 226.5 (236.37)
  WEEK 10 ; 4 to 8 HOURS POST-DOSE; n=13, 13, 11: number analyzed (Participants) | 13 | 13 | 11
  WEEK 10 ; 4 to 8 HOURS POST-DOSE; n=13, 13, 11 | 92.6 (169.45) | 81.8 (168.16) | 429.2 (735.69)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-SAEs were collected from the start of the study treatment up to 3.2 years.
Description: On-treatment SAEs and non-SAEs were collected in Safety Population which included all the participants who received at least one dose of randomized treatment and was based on the actual treatment received.
Arm/Group | Dabrafenib Followed by Combination Therapy | Trametinib Followed by Combination Therapy | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/16 | 2/16
Serious Adverse Events (participants affected / at risk) | 8/16 | 7/16 | 4/16
Other Adverse Events (participants affected / at risk) | 16/16 | 16/16 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabrafenib Followed by Combination Therapy (N=16) | Trametinib Followed by Combination Therapy (N=16) | Combination Therapy (N=16)
Pyrexia (General disorders) | 2 (3) | 3 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabrafenib Followed by Combination Therapy (N=16) | Trametinib Followed by Combination Therapy (N=16) | Combination Therapy (N=16)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (14) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 2 (3)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Histiocytosis Haematophagic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tricuspid Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 2 (3) | 1 (2) | 2 (2)
Eye Pain (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 7 (19) | 5 (7)
Nausea (Gastrointestinal disorders) | 8 (12) | 4 (11) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (6) | 4 (9) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (6) | 5 (6) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (4) | 2 (6) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (4) | 4 (5) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (3) | 4 (4) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Aerophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Painful Defaecation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tooth Demineralisation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth Discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal Fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue Discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (12) | 13 (49) | 6 (18)
Hyperthermia (General disorders) | 4 (13) | 4 (15) | 4 (22)
Asthenia (General disorders) | 10 (14) | 10 (20) | 9 (17)
Chills (General disorders) | 3 (4) | 10 (15) | 4 (8)
Oedema Peripheral (General disorders) | 4 (7) | 6 (8) | 4 (4)
Chest Pain (General disorders) | 3 (6) | 1 (2) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 4 (4) | 1 (1)
Influenza Like Illness (General disorders) | 3 (3) | 2 (2) | 3 (3)
Xerosis (General disorders) | 3 (3) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling Of Body Temperature Change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-Defined Disorder (General disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammatory Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal Dryness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema Due To Cardiac Disease (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1) | 3 (3) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy To Arthropod Sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 7 (8) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 4 (4) | 3 (4)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Rash Pustular (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Molluscum Contagiosum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Fungal Oesophagitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Moraxella Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 5 (15) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 5 (14) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 2 (10) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 5 (8) | 7 (9) | 5 (7)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 2 (7) | 0 (0)
Lipase Increased (Investigations) | 1 (2) | 2 (4) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 2 (3) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Ejection Fraction Decreased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 1 (3) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 1 (2) | 1 (1)
Amylase Increased (Investigations) | 0 (0) | 1 (2) | 1 (1)
Blood Triglycerides Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Intraocular Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Albumin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Fibrinogen Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (7) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Weight Fluctuation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (5) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 (7) | 6 (9) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (8) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (8) | 4 (7)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (7) | 5 (7) | 3 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (6) | 2 (3)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (5) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (16) | 9 (15) | 6 (9)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 3 (7)
Paraesthesia (Nervous system disorders) | 2 (5) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Burning Sensation (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (2)
Cervical Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine With Aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Demyelinating Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Head Discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Contractions Involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood Altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Tubular Acidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 8 (15) | 3 (3)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6 (9) | 2 (3) | 1 (1)
Palmoplantar Keratoderma (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6) | 6 (7) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (7) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (5)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 2 (2)
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 2 (3)
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophilic Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot Flush (Vascular disorders) | 1 (3) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (3) | 2 (3) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Venous Disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2013-10-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT02314143/Prot_000.pdf
  • Statistical Analysis Plan (2015-01-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT02314143/SAP_001.pdf